CLINICAL TRIAL: NCT02312895
Title: Randomized Controlled Trial Comparing the Use of Dry Needling to Manual Therapy for Patients With Mechanical Low Back Pain.
Brief Title: Comparing Dry Needling to Manual Therapy for Patients With Mechanical Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 159-14
Record Dates: First submitted 2014-11-24; First posted 2014-12-09 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling (Experimental): A total of 30 subjects will be randomized to this experimental arm. If randomized to this arm, subjects will receive dry needling, patient education, and a home exercise program.
  Interventions: Other: Dry needling; Other: Home Exercise Program
- Manual Therapy (Experimental): A total of 30 subjects will be randomized to this experimental arm. If randomized to this arm, subjects will receive manual therapy, patient education, and a home exercise program.
  Interventions: Other: Manual therapy; Other: Home Exercise Program

INTERVENTIONS:
Other: Manual therapy — The therapist will locate the involved segment using passive accessory intervertebral movements. The segment will be localized to the level, which provokes the patient's symptoms most easily, and this segment will be determined to be the involved level. Once this level has been identified, the therapist will compare central glides over the spinous process or a unilateral glide over the facet joint to determine which is more provocative. Whichever is most provocative will be the location of the treatment. The therapist will provide 3 bouts lasting 45 seconds just easing into the patient's symptoms at the most provocative level with approximately 45 seconds rest between each bout.
  Arms: Manual Therapy
Other: Dry needling — Dry needling involves inserting a dry, mono-filament needle through the skin and into an area of symptomatic soft tissue. The two-inch needles will be placed segmentally and into the lower extremities following peripheral nerve patterning by the treating physical therapist. Following initial penetration into the skin over the tender area, the therapist carefully advances the needle into the tissue below the skin. After the needle has reached the desired depth, the therapist will insert the subsequent needles. Needles will be placed along the segmental levels of the lumbar spine above and below the tender area identified and into the lower extremity in areas that correlate with a peripheral nerve map. Needles will remain in the tissue for up to 5 minutes, removed, and appropriately disposed of.
  Arms: Dry Needling
Other: Home Exercise Program — A home exercise program will be given to each subject to be completed in the clinic and at home 1x/day. The exercises will consist of active range of motion exercises and core stabilization exercises. The program is standardized for all subjects.

SUMMARY:
This is a comparative study to determine if there is a difference in pain reduction and disability between dry needling and manual therapy for patients with low back pain. Subjects will be seen two times per week for 3 weeks (6 visits) and will receive either dry needling or manual mobilizations along with patient education and a home exercise program.

DETAILED DESCRIPTION:
Procedures:

Subjects will sign the informed consent prior to any examination procedures. Eligibility assessment will be performed by the treating physical therapist and will include the subject filling out the demographic / health history questionnaire, outcome measures, and a clinical examination. The treating physical therapist will use 2 components of the examination for eligibility criteria into the study. The treating therapist will press on the subject's joints in their back to try to elicit their chief complaint. The treating physical therapist will also press on the soft tissue of the subject's back to check for any symptomatic points. A symptomatic point would include recreation of their chief complaint, tenderness, hypersensitivity, or referred pain. The treating physical therapist will then draw an X on the patient's back where the most symptomatic tissue exists. This point will be used by the data collecting physical therapist in order to collect pain pressure threshold of the area.

The data collecting physical therapist will have the subject complete an Oswestry Disability Index(ODI), gather a measure of the pain from the patient ,and the pain pressure threshold. Each subject will then be allocated to either the manual therapy group or the dry needling group.

Once a subject is assigned to a group, they will receive either dry needling or manual therapy mobilizations by the treating therapist. Each subject will remain in the assigned group as long as they are continuing in the study up to 3 weeks. In addition to the treatments under investigation, a standardized home exercise program will be assigned to each of the subjects by the treating physical therapist. This program will be given to and reviewed with each subject to ensure they understand the exercises and will perform the exercise program 1x/day for the duration they are under the care of the physical therapist for the study. Subjects will be treated on day 1 of their plan of care and subsequent treatments will occur 2x/week for a total of 3 weeks, unless discharge occurs earlier than the 3 week data point. Early discharge will occur if the subject achieves resolution of symptoms or if they decide they no longer wish to be a research participant.

Subsequent sessions will involve the collection of outcome data by the data-collecting therapist followed by treatment performed by the treating physical therapist. No adjustments will be made to the treatment protocol in any of the sessions. Subjects will only be scheduled with and treated by the same treating physical therapist each session. In the event that a treating physical therapist is unable to see a subject participating in the study, the subject will be rescheduled for a different time to receive care.

ELIGIBILITY:
Inclusion Criteria:

* There will be 72 subjects participating in this study that present with mechanical low back pain, ranging from 18-70 years old. The 72 subjects includes a 20% attrition rate 12 additional subjects. The total needed for analysis is 60 subjects, 30 per group.

Exclusion Criteria:

* Subjects will be excluded if the examining therapist cannot provoke either active or latent MTrPs of the subject's low back muscles and/or elicit symptoms with manual passive movement of the spine at the joints of the low back. Exclusion criteria will also consist of the presence of any red flags revealed in the patient history (i.e., tumor, metabolic diseases, RA, osteoporosis, prolonged history of steroid use, prior lumbar surgery, current pregnancy, etc.) or examination (i.e. signs consistent with significant nerve root compression). Subjects will be excluded if they demonstrate signs of Chronic Regional Pain Syndrome (CRPS), are currently seeking litigation, are unable to speak English, and/or have been diagnosed with a condition that can cause prolonged MTrPs such as fibromyalgia, hypothyroidism, or iron deficiency. In addition, no patients who have a transmittable blood disease will be included.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (change over time) | The ODI will be recorded at baseline, 1 week, 2 weeks, and discharge/3 weeks.
  The ODI is a ten question self report measure that assesses the impact of the patient's pain on their ability to perform everyday activities and is currently considered the gold standard for measuring degree of disability and estimating quality of life in a person with low back pain.

SECONDARY OUTCOMES:
Numerical Pain Rating Scale (change over time) | The NPRS will be recorded at baseline, immediately following treatment, at 1 week, 2 weeks, and discharge/3 weeks.
  The patient is asked to rate their level of pain on an 11-point numerical scale 0-10 with 0 being "no pain" and 10 being the "worst possible pain." Pain will be recorded one additional time after the initial treatment session.
Pain pressure threshold (change over time) | The NPRS will be recorded at baseline, immediately following treatment, at 1 week, 2 weeks, and discharge/3 weeks.
  PPT will be measured as described above using an algometer to the identified MTrPs. An algometer is an instrument that detects sensitivity to pressure. The force gauge algometer is placed on the area of a patient's identified MTrP. Pressure is gradually increased until the person perceives a noxious sensation. The amount of pressure at the point of pain is recorded then repeated and and PPT will be performed twice each time, and the measures will be averaged together for data analysis. PPT will be collected one additional time post treatment session 1.
Percentage of recovery (one time assessment at the end of the 3 weeks) | 3 weeks or Discharge
  A global percentage of improvement is a measure of the patient's perception of the change in their condition. It will be recorded at discharge by asking the subject what percent better they believe their low back problem is compared to when they entered the study.
Patient Specific Functional Scale Score | PSFS score collected at baseline, 1 week, 2 weeks, and 3 weeks or discharge
  The PSFS is a patient identified self-report questionnaire that measures general activity limitations. The scale ranges from 0 (unable to perform) to 10 (able to perform the activity at the level prior to injury). The patient reports 3 activities and rates each activity from 0 to 10, which are averaged for a composite score.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Learman, PhD, Principal Investigator — Faculty; David W Griswold, Doctorate, Principal Investigator — Faculty
Locations (1):
- Youngstown state university, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Furlan AD, van Tulder M, Cherkin D, Tsukayama H, Lao L, Koes B, Berman B. Acupuncture and dry-needling for low back pain: an updated systematic review within the framework of the cochrane collaboration. Spine (Phila Pa 1976). 2005 Apr 15;30(8):944-63. doi: 10.1097/01.brs.0000158941.21571.01. PMID 15834340
- [Background] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800
- [Background] Cook C, Learman K, Showalter C, Kabbaz V, O'Halloran B. Early use of thrust manipulation versus non-thrust manipulation: a randomized clinical trial. Man Ther. 2013 Jun;18(3):191-8. doi: 10.1016/j.math.2012.08.005. Epub 2012 Oct 2. PMID 23040656